CLINICAL TRIAL: NCT05327556
Title: Epinephrine in the Pediatric Intensive Care Unit: A Dose-Effect Trial (EPI Dose)
Brief Title: Epinephrine in the Pediatric Intensive Care Unit: A Dose-Effect Trial
Acronym: EPIDose
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding constraints
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Catherine E. Ross, MD, Attending Physician, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P00035730
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study kits in either arm will be identical, and only the research pharmacy and the study statisticians will have access to the populated Master Randomization List.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.5 mcg/kg Dose (Active Comparator): Providers use 0.1 mL/kg of 5 mcg/mL epinephrine for target dose 0.5 mcg/kg
  Interventions: Drug: Epinephrine 0.5 mcg/kg
- 1.0 mcg/kg Dose (Active Comparator): Providers use 0.1 mL/kg of 10 mcg/mL epinephrine for target dose of 1.0 mcg/kg
  Interventions: Drug: Epinephrine 1 mcg/kg

INTERVENTIONS:
Drug: Epinephrine 0.5 mcg/kg — Syringe with 5 mcg/mL epinephrine
  Other Names: Peri-Arrest Bolus Epinephrine
  Arms: 0.5 mcg/kg Dose
Drug: Epinephrine 1 mcg/kg — Syringe with 10 mcg/mL epinephrine
  Other Names: Peri-Arrest Bolus Epinephrine
  Arms: 1.0 mcg/kg Dose

SUMMARY:
The use of peri-arrest bolus epinephrine (PBE) has emerged as a rescue strategy for life-threatening hypotension in pediatric intensive care units (ICU) despite scant published data supporting its use in this setting. As optimal dosing of PBE in this population is unclear, we aim to determine if an initial dose of 0.5 mcg/kg versus 1.0 mcg/kg yields differences in hemodynamic outcomes. The EPI Dose Study is a single-center, prospective, randomized, double-blind, dose-effect trial measuring systolic blood pressure (SBP) before and after PBE is given. We hypothesize that the 1.0 mcg/kg group will have more robust increases in SBP.

DETAILED DESCRIPTION:
In order to test the hypothesis that PBE doses of 1.0 mcg/kg will have more robust increases in SBP as compared to 0.5 mcg/kg in critically ill children and young adults with acute hypotension, we plan to conduct a Phase II, single-center, prospective, randomized, double-blind, dose-effect trial. Children and young adults <26 years of age who, at the discretion of the clinical team, require rescue PBE for life-threatening hypotension and meet inclusion/exclusion criteria will be enrolled. Prior to randomization, our pharmacy team will prepare treatment packets with 3 pre-mixed PBE which will be stocked in the ICUs with either 5 mcg/mL or 10 mcg/mL of epinephrine. Clinicians will be instructed to use 0.1 mL/kg of the experimental syringe for the initial dose, resulting in target doses of 0.5 mcg/kg (Arm 1) or 1 mcg/kg (Arm 2), respectively. Treatment packs will be labeled according to the randomization scheme, and only the pharmacy team will have knowledge of the concentration of epinephrine in each package. Nurses will be instructed to record the exact time of the experimental dose, around which all time-sensitive data will be collected. The clinicians, patients and research team will be blinded to the intervention. We will not restrict any other interventions chosen by the clinical team. Unblinded interim analyses will be performed after the first 6 months of enrollment, and every 12 months thereafter through study completion and reported to the Data and Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female less than 26 years of age.
2. Admitted to BCH and receiving care in a participating ICU.
3. Is prescribed BDE for acute hypotension deemed to be life-threatening in the judgement of the treating clinician.

Exclusion Criteria:

1. Has opted out of the study prior to enrollment.
2. Has orders in place which limit resuscitation efforts.
3. Is actively receiving chest compressions while PBE is administered.
4. Is receiving care in the neonatal intensive care unit.
5. Is receiving care outside of the ICU at the time PBE is administered (i.e procedural areas).
6. Is pregnant or breastfeeding.
7. Is a prisoner.
8. Is a ward if the state (DCF custody).

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | 10 minutes
  The lowest systolic blood pressure value in the 5 minutes prior to or up to 1 minute after the documented time of PBE administration (nadir) subtracted from the highest systolic blood pressure in the 5 minutes following PBE (must be subsequent to the nadir). If an additional dose of PBE was administered within 5 minutes of the initial dose, the peak SBP will be the highest value recorded prior to the subsequent dose.
  Primary analysis will be performed with an intention-to-treat approach based on the concentration of study drug received. An exploratory analysis will be performed per protocol based on the actual volume of study drug the patient received on first administration being within 20% of the intended volume. Patients who received ≥0.4 to ≤0.6 mcg/kg will be considered in the 0.5 mcg/kg group whereas patients who received ≥0.8 to ≤1.2 mcg/kg will be considered in the 1 mcg/kg group.

SECONDARY OUTCOMES:
Incidence of Severe (Stage II) Hypertension | 5 minutes
  The proportion of patients whose peak systolic blood pressure (determined as per the primary outcome) is greater than or equal to the 95th percentile plus 12 mmHg or greater than or equal to 140 mmHg, whichever is lower.

OTHER OUTCOMES:
Incidence of Cardiac Arrest | 0 to 120 minutes
  The proportion of patients who receive chest compressions at anytime from 0 to 120 minutes after the first dose of study drug
Incidence of Extra-corporeal Membrane Oxygenation (ECMO) | 0 to 120 minutes
  The proportion of patients who are cannulated to ECMO at anytime from 0 to 120 minutes after the first dose of study drug, starting at time of first flow
Early Survival | 7 days
  The proportion of patients alive or discharged from the hospital alive at 7 days after the calendar day study drug was administered
Survival to Hospital Discharge | 90 days
  The proportion of patients alive at time of discharge from the hospital (Truncated at 90 days)
Change in Heart Rate (HR) | 10 minutes
  Difference in HR before and after PBE is given, using measurements that coincide with the primary outcome
Change in Mean Arterial Pressure (MAP) | 10 minutes
  Difference in MAP before and after PBE is given, using measurements that coincide with the primary outcome
Change in Diastolic Blood Pressure (DBP) | 10 minutes
  Difference in DBP before and after PBE is given, using measurements that coincide with the primary outcome
Percent Change in Vital Signs | 10 minutes
  The difference in SBP, MAP, DBP and HR (defined as above) expressed as a percentage.
Incidence of Stage I Hypertension (or greater) | 5 minutes
  The proportion of patients whose peak systolic blood pressure (as per the primary outcome) is greater than or equal to the 95th percentile or 130/80 mm Hg (whichever is lower).
Incidence of Extreme Hypertension | 5 minutes
  The proportion of patients whose peak systolic blood pressure (as per the primary outcome) is greater than or equal to the 95th percentile + 30 mm Hg or ≥170, whichever is lower.
Incidence of Non-Responders | 10 minutes
  The proportion of patients who do not respond to initial dose of study drug, defined as <10mmHg difference between nadir and peak SBP
Number of doses of epinephrine per resuscitation episode | 120 minutes
  Comparison of the number of doses of epinephrine (study drug or open label) given in a discrete resuscitation episode up to 120 minutes after initial dose.
Total dose of epinephrine per resuscitation episode | 120 minutes
  Comparison of the total dose of epinephrine (study drug or open label) in mcg/kg given in a discrete resuscitation episode up to 120 minutes after initial dose.
Safety Outcomes | 0 to 7 days
  The proportion of patients who develop the following prespecified safety outcomes:
  * Any new arrhythmia within 20 minutes of first dose of study drug
  * Any new arrhythmia requiring intervention within 20 minutes of first dose of study drug
  * Intracranial hemorrhage associated with severe or extreme hypertension within 5 minutes of the first dose of study drug which is diagnosed within 7 days after the calendar day study drug was administered
Continuous Dose Effect Curve | 10 minutes
  Correlation of actual dose received in mcg/kg with change in systolic blood pressure.
Effect on change in Systolic Blood Pressure by treatment group | 10 minutes
  Effect on change in Systolic Blood Pressure by treatment group controlling for:
  * Age
  * Nadir BP adjusted for age per PALS handbook (≤28 days of age, SBP <60 mmHg; ≥29 days to <1 year, SBP <70 mmHg; ≥1 year to <10 years, SBP <70 + 2x(age in years) mmHg; and ≥10 years, SBP <90 mmHg.)
  * Provider who was leading the event

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Ross, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified individual participant data collected during the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication of primary results and ending 5 years after publication.
Access Criteria: Data will be made available on a case by case basis to investigators whose proposed use of the data has been approved by the primary investigator.

REFERENCES:
- [Background] Ross CE, Asaro LA, Wypij D, Holland CC, Donnino MW, Kleinman ME. Physiologic response to pre-arrest bolus dilute epinephrine in the pediatric intensive care unit. Resuscitation. 2018 May;126:137-142. doi: 10.1016/j.resuscitation.2018.03.011. Epub 2018 Mar 8. PMID 29526678